CLINICAL TRIAL: NCT03319966
Title: Eyetracking and Neurovision Rehabilitation of Oculomotor Dysfunction in Mild Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HSR#17-4409
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Mild Traumatic Brain Injury; Brain Concussion; Convergence Insufficiency; Accommodative Insufficiency; Saccadic Eye Movement Deficiency; Oculomotor Dysfunction
MeSH Terms: conditions — Brain Concussion; Ocular Motility Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oculomotor Dysfunction: This group consists of subjects with mTBI who have been diagnosed with OMD by objective OD measurements. These subjects will undergo neurovision rehabilitation used to treat oculomotor dysfunction following traumatic brain injury per usual clinical standard of care at the HCMC TBI Clinic.

SUMMARY:
The purpose of this single center, longitudinal, pilot study is to provide evidence for the use of an eye tracking system as an objective tool to identify mild traumatic brain injury (mTBI) related oculomotor dysfunction (OMD) and predict the effectiveness of neurovision rehabilitation (NVR) of OMD. Eye tracking visual stimulus measurements will be compared to objective developmental optometrist (OD) diagnosis and assessments. It will be determined whether an eye tracking system can predict the presence or absence of mTBI related OMD and whether mTBI patients who have OMD based on the eye tracking system will respond positively to NVR.

DETAILED DESCRIPTION:
The primary objectives are: 1) To demonstrate that measurements from visual stimulus and eye tracking system will predict the presence or absence of traumatic brain injury related vision disorder, i.e. oculomotor dysfunction (OMD) as diagnosed by a developmental optometrist (OD). 2) To use the eye tracking visual measurements to predict the effectiveness of neurovision rehabilitation (NVR) on post-traumatic OMD by comparing the data obtained to the objective visual measurements found on the OD examination.

Mild traumatic brain injury (mTBI) that alters brain function is a major public health concern of significant personal and societal burden. Mild traumatic brain injury patients may experience any or all of at least 20 symptoms, with some persisting for weeks to months and increasing the risk of comorbidities. Current mTBI diagnosis and treatment are subjective and imprecise rather than objective and patient specific. Despite the varied heterogeneous manifestations of mTBI based on location and severity of injury as well as predisposing factors, treatment is generic and lacking in active therapies: rest with the avoidance of devices/screens to avoid exacerbating symptoms. This "one size fits all" approach is suboptimal, often resulting in ineffective management with prolonged inadequate recovery. Recent evidence suggests effective therapies to be specific to the mTBI patient and their symptoms with promising interventions targeting vestibular deficits as well as post-TBI OMD NVR. Neurovision rehabilitation is analogous to physical therapy for the eyes and improves the connection between the brain and the eyes with prior research finding NVR to be very effective for patients with post-concussion visual dysfunctions. Patients with potential mTBI primarily present to the emergency department, primary care, or specialty clinic, where there lacks proper equipment, training, and time for a comprehensive vision examination. Additionally, identification and diagnosis of OMD is only conducted currently by a vision specialist or highly skilled TBI specialists. This leaves a majority of OMD patients with inappropriate diagnosis and inadequate work or school accommodations as well as without treatment with NVR, lenses, and prisms. Thus an objective, easily accessible tool to identify mTBI related OMD would greatly advance clinical care.

This trial is a single center, longitudinal, pilot study. One hundred mTBI patients with OMD, confirmed with objective testing by a OD, who fit inclusion/exclusion criteria will be initially identified by providers at the Hennepin County Medical Center (HCMC) TBI Clinic. No subject will be excluded on the basis of sex/gender, race or ethnicity. If interested, subjects will be consented then undergo an initial eye tracking. Within two weeks of the initial eye tracking, subjects will begin recommended NVR with occupational therapists (OT) at HCMC. Each NVR session will assess each subject's progress and following each NVR session, subjects will receive an eye tracking test. Additionally, within two months of the initial OMD diagnosis patients will follow up with the OD every two months until their OMD is resolved or until one year following their diagnosis. Subjects will also undergo an eye tracking test after each OD follow up appointment. Eye tracking visual stimulus measurements will be compared to OD diagnostic measurements and assessments.

The goals of this research study are to improve objective, timely identification of mTBI related visual dysfunctions and assessment of the effectiveness of NVR. A positive outcome will greatly impact diagnosis and care of mTBI patients with vision dysfunction, as objective assessments will be more widely and readily available and NVR will be more utilized by the medical community. Overall post-mTBI functional outcomes will improve, significantly lessening this major public health concern affecting patients, families, communities, and society.

ELIGIBILITY:
Inclusion Criteria:

* Mild traumatic brain injury (Glasgow Coma Scale ≥ 13)
* Post traumatic amnesia < 24 hours
* Diagnosed with oculomotor dysfunction by developmental optometrist and neurovision rehabilitation recommended
* Time of traumatic brain injury ≤ 2 years
* Informed consent obtained

Exclusion Criteria:

* Glasgow Coma Scale < 13
* Age < 13 years and > 55 years
* Time of traumatic brain injury > 2 years
* Cranial nerve II, III, IV, or VI palsy
* History of strabismus
* Monocular vision, including Lasik surgery for monofixation
* Taking medications known to interfere with visual process/recovery
* Taking illicit drugs such as marijuana, cocaine, heroin, etc.

Ages: 13 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Mild traumatic brain injury patients who meet the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
Eye Tracker as an Objective Tool for "Yes/No" Assessment of Oculomotor Dysfunction Presence | 12 months
  Eye tracker metrics of oculomotor dysfunction as compared to objective developmental optometry diagnostic measurements.

SECONDARY OUTCOMES:
Eye Tracking Visual Measurements as Objective Predictor of Neurovision Rehabilitation Effectiveness | 12 months
  Eye tracker metrics of oculomotor dysfunction status throughout neurovision rehabilitation as compared to objective developmental optometry follow up measurements and eye therapy exercise findings.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Rockswold, MD, Principal Investigator — Hennepin County Medical Center, Minneapolis
Locations (1):
- Hennepin County Medical Center Traumatic Brain Injury Clinic, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided